CLINICAL TRIAL: NCT00232505
Title: Phase II Trial of Cetuximab Alone and in Combination With Carboplatin in ER-Negative, PR-Negative, HER-2 Nonoverexpressing Metastatic Breast Cancer
Brief Title: Cetuximab + / - Carboplatin for Estrogen Receptor-Negative, Progesterone Receptor-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bristol-Myers Squibb (Industry); Avon Foundation (Other); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LCCC 0403; M01RR000046 (NIH); CA058223 (Other Grant/Funding Number: NCI OSP/SPOREs); NCT00420329 (obsolete NCT alias); NCT00492375 (obsolete NCT alias)
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cetuximab; Carboplatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab (Experimental): Patients receive cetuximab IV over 60-120 minutes once a week. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients not responding to treatment may cross over to arm II.
  Interventions: Biological: cetuximab
- Cetuximab and Carboplatin (Experimental): Patients receive cetuximab as in arm I and carboplatin IV on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: carboplatin

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: Erbitux
Drug: carboplatin — Given IV
  Other Names: Paraplatin
  Arms: Cetuximab and Carboplatin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Cetuximab may also stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving cetuximab together with carboplatin is more effective than giving cetuximab alone in treating metastatic breast cancer.

PURPOSE: This randomized phase II trial is studying cetuximab and carboplatin to see how well they work compared with cetuximab alone in treating women with estrogen receptor-negative (ER-), progesterone receptor-negative (PR-) metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall response rate in women with estrogen receptor-negative, progesterone receptor-negative, human epidermal growth factor receptor 2 (HER2)-nonoverexpressing metastatic breast cancer treated with cetuximab with vs without carboplatin.

Secondary

* Compare the time to disease progression in patients treated with these regimens.
* Correlate downstream effects of epidermal growth factor receptor (EGFR) inhibitor on Mitogen-activated protein kinases (MAPK), Protein kinase B (AKT), monoclonal antibody Ki-67 (Ki67), and EGFR-dependent signaling, proliferation, and apoptosis with toxicity and response in patients with accessible tumors treated with these regimens.
* Determine the changes in biomarkers and gene expression in circulating tumor cells during treatment.
* Compare the overall survival rate in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive cetuximab IV over 60-120 minutes once a week.
* Arm II: Patients receive cetuximab as in arm I and carboplatin IV on days 1, 8, and 15.

In both arms, treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients not responding to treatment in arm I may cross over to arm II.

Blood samples are collected periodically throughout study for correlative biomarker analysis by Immunohistochemistry (IHC) and gene expression analysis.

After completion of study treatment, patients are followed every 4 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Metastatic (stage IV) disease
* Measurable disease by RECIST criteria

  * Irradiated lesions are not considered measurable disease
* Central nervous system (CNS) metastases allowed if disease is stable (no evidence of progression) ≥ 3 months after local therapy
* No lesions identifiable only by positron emission tomography (PET) scan
* HER2 nonoverexpressing disease by IHC (0 or 1) or non-gene amplified by Fluorescence In Situ Hybridization (FISH)

  * HER2 2+ by IHC allowed
* Hormone receptor status:

  * Estrogen receptor-negative and progesterone receptor-negative tumor

Inclusion Criteria

* At least 18 years of age
* Metastatic breast cancer (Stage IV) with measurable disease by RECIST criteria
* No more than three prior chemotherapy regimens either in the adjuvant or metastatic setting.
* Histologically documented (either primary or metastatic site) breast cancer that is estrogen receptor- (ER-) negative, PR-negative, and HER-2 nonoverexpressing by immunohistochemistry (0,1) or non-gene amplified by FISH performed upon the primary tumor or metastatic lesion. HER-2 2+ by immunohistochemistry is usually negative by FISH, and this confirmatory test should be performed when possible, however may participate if fulfill other criteria.
* Completion of prior chemotherapy at least 3 weeks prior to study entry.
* Patients may have received therapy (ies) in the adjuvant or metastatic setting, however must have discontinued prior to entry. Patients may receive concurrent bisphosphonates, however if taking bisphosphonates, bone lesions may not be used for progression or response.
* Radiation therapy must be completed at least 2 weeks prior to study entry, and radiated lesions may not serve as measurable disease.
* Patients may have CNS metastases if stable (no evidence of progression) > 3 months after local therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2 and life expectancy of at least 6 months.
* Adequate organ function defined as:absolute neutrophil count (ANC) > 1500/mm3, plts > 100,000/mm3, creatinine clearance >50 mL/min, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN) (or ≤5 x ULN in case of liver metastases); total bilirubin ≤1.5 mg/dL.
* Tissue block available for EGFR studies is recommended, although will not exclude patients from participating.
* Pregnant or lactating women will be excluded. Women of child bearing potential must have documented negative pregnancy test within two weeks of study entry and agree to acceptable birth control during the duration of the study therapy.
* Signed written informed consent.

Exclusion Criteria

* Lesions identifiable only by PET.
* More than three prior chemotherapy regimens (including adjuvant). Sequential regimens such as doxorubicin and cyclophosphamide followed by paclitaxel (AC-paclitaxel) are considered one regimen.
* Prior therapy which specifically and directly targets the EGFR pathway with therapeutic intent.
* Prior platinum agent for metastatic disease. If platinum agent was used adjuvantly, the patient must have had at least 12 months disease-free interval prior to relapse.
* Prior severe infusion reaction to a monoclonal antibody.
* Major medical conditions that might affect study participation (uncontrolled pulmonary, renal, or hepatic dysfunction, uncontrolled infection).
* Significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy that is either symptomatic or asymptomatic but with decreased ejection fraction <45%
* Other significant comorbid condition which the investigator feels might compromise effective and safe participation in the study.
* Inability to comply with the requirements of the study.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-11 (Actual); Primary Completion 2010-06-21 (Actual); Study Completion 2012-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Carey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (14):
- United States (14):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carey LA, Rugo HS, Marcom PK, Mayer EL, Esteva FJ, Ma CX, Liu MC, Storniolo AM, Rimawi MF, Forero-Torres A, Wolff AC, Hobday TJ, Ivanova A, Chiu WK, Ferraro M, Burrows E, Bernard PS, Hoadley KA, Perou CM, Winer EP. TBCRC 001: randomized phase II study of cetuximab in combination with carboplatin in stage IV triple-negative breast cancer. J Clin Oncol. 2012 Jul 20;30(21):2615-23. doi: 10.1200/JCO.2010.34.5579. Epub 2012 Jun 4. PMID 22665533
- [Derived] Oliveras-Ferraros C, Vazquez-Martin A, Lopez-Bonet E, Martin-Castillo B, Del Barco S, Brunet J, Menendez JA. Growth and molecular interactions of the anti-EGFR antibody cetuximab and the DNA cross-linking agent cisplatin in gefitinib-resistant MDA-MB-468 cells: new prospects in the treatment of triple-negative/basal-like breast cancer. Int J Oncol. 2008 Dec;33(6):1165-76. PMID 19020749
- See also: University of North Carolina Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between December 2005 and October 2007 from thirteen cancer centers throughout the US.
Pre-assignment Details: Four patients declined participation for personal reasons, three were screen failures, three had death or progression during the screening period.
Period: Overall Study
Arm/Group | Cetuximab | Cetuximab and Carboplatin
Started | 31 | 71
Not Evaluable | 0 | 6
Early Progressors | 2 | 5
Off Protocol | 5 | 0
Completed | 26 | 60
Not Completed | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab | Cetuximab and Carboplatin | Total
Number analyzed (Participants) | 31 | 71 | 102
Age, Continuous [Median (Full Range); unit: years] | 49 [33 to 71] | 52 [28 to 83] | 50.5 [28 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 71 | 102
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 17 | 28
  White | 19 | 51 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 71 | 102
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — A scale from 0-5 to describe a patient's level of functioning in terms of selfcare ability and activity level.
  0, Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 17 | 37 | 54
    1 | 14 | 28 | 42
    2 | 0 | 4 | 4
    missing | 0 | 2 | 2
Menopausal Status [Count of Participants; unit: Participants]
  Postmenopausal | 21 | 56 | 77
  Pre- or perimenopausal | 10 | 15 | 25
Dominant metastatic site [Count of Participants; unit: Participants]
  Lung | 9 | 20 | 29
  Liver | 8 | 17 | 25
  Lymph nodes | 4 | 14 | 18
  Locoregional | 5 | 10 | 15
  Bone | 1 | 4 | 5
  Skin/soft tissue | 3 | 5 | 8
  Other | 1 | 1 | 2
Treatment [Number; unit: participants]
  Prior chemotherapy | 30 | 67 | 97
  Adjuvant/neoadjuvant | 26 | 60 | 86
  Metastatic | 21 | 34 | 55

OUTCOME MEASURES:

1. Primary Outcome: Overall Disease Response Rate
Description: Overall response rate of single agent cetuximab and cetuximab + carboplatin will be measured by radiographic response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria every 8 weeks until subject experiences disease progression. Overall response will be measured as complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD).Per RECIST v1.0 for target lesions and assessed by CT (spiral): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Cetuximab and Carboplatin After Cetuximab Alone: Patients from Arm 1 who progressed on cetuximab alone who went on to receive cetuximab + carboplatin
- Cetuximab and Carboplatin Subset: patients receiving cetuximab and carboplatin who had confirmed basal-like disease by quantitative realtime polymerase chain reaction-based intrinsic subtype assay
Arm/Group | Cetuximab | Cetuximab and Carboplatin After Cetuximab Alone | Cetuximab and Carboplatin | Cetuximab and Carboplatin Subset
Number analyzed (Participants) | 31 | 25 | 71 | 51
Participants
  Complete response | 0 | 0 | 1 | 1
  Partial response | 2 | 4 | 11 | 17
  Stable disease | 3 | 7 | 15 | 8
  Stable disease > 6 months | 1 | 3 | 10 | 7
  Progressive disease | 26 | 12 | 38 | 32
  Not evaluable | 0 | 2 | 6 | 3

2. Secondary Outcome: Overall Survival
Description: Subjects will be contacted every 4 months after discontinuation of active treatment to assess survival.
Time Frame: Every four months until death of any cause or end of data collection up to 40 months
Measure: Number; unit: participants surviving
Arm/Group | Cetuximab | Cetuximab and Carboplatin
Number analyzed (Participants) | 31 | 71
participants surviving
  Baseline | 31 | 71
  4 months | 22 | 56
  8 months | 12 | 41
  12 months | 9 | 30
  16 months | 8 | 23
  20 months | 8 | 19
  24 months | 6 | 8
  28 months | 5 | 4
  32 months | 1 | 3
  36 months | 1 | 2
  40 months | 0 | 0

3. Secondary Outcome: Progression-Free Survival
Description: Time to disease progression of cetuximab or cetuximab + carboplatin as indicated by radiographic assessment
Time Frame: Every four months until progression, death of any cause, or end of data collection up to 40 months
Measure: Number; unit: participants
Arm/Group | Cetuximab | Cetuximab and Carboplatin
Number analyzed (Participants) | 31 | 71
participants
  Baseline | 31 | 71
  4 months | 4 | 27
  8 months | 2 | 11
  12 months | 2 | 7
  16 months | 1 | 7
  20 months | 1 | 6
  24 months | 1 | 6
  28 months | 1 | 1
  32 months | 1 | 1
  36 months | 1 | 1
  40 months | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 30 days after treatment
Description: Categorical "Other, Specify" events listed below include verbatim from data collection source in footnotes
Arm/Group | Cetuximab | Cetuximab and Carboplatin After Cetuximab Alone | Cetuximab and Carboplatin
Serious Adverse Events (participants affected / at risk) | 3/31 | 8/25 | 20/71
Other Adverse Events (participants affected / at risk) | 27/31 | 24/25 | 68/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=31) | Cetuximab and Carboplatin After Cetuximab Alone (N=25) | Cetuximab and Carboplatin (N=71)
Edema: limb (Blood and lymphatic system disorders) | 2 | 1 | 0
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 | 3 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1
Cardiac General - Other (Specify, __) (Cardiac disorders) | 0 | 1 | 0 — tachycardia
Cardiac General - Other (Specify, __) (Cardiac disorders) | 0 | 0 | 1 — Port fracture: tubing embolized to main pulm artery
Confusion (Psychiatric disorders) | 0 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7
Extremity-lower (gait/walking) (General disorders) | 0 | 0 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 | 1 | 1
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 2
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 1 | 0 | 0 — abdomen swelling, distension
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 0 | 1 | 0 — hepatic encephalopathy
Hemorrhage, CNS (Nervous system disorders) | 0 | 0 | 1
Hemorrhage, GI - Esophagus (Gastrointestinal disorders) | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (ANC <1.0 x 10e (Infections and infestations) | 0 | 1 | 0 — Wound
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 0 | 1 | 0
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 2
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 0 | 0 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 1 | 1
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain - Chest/thorax NOS (General disorders) | 0 | 0 | 2
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain - Middle ear (Ear and labyrinth disorders) | 0 | 1 | 0
Pain - Other (Specify, __) (General disorders) | 0 | 1 | 0 — intolerable pain in sternum
Pain - Other (Specify, __) (General disorders) | 0 | 2 | 0 — pain in arm due to lymphedema
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 0 | 3
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 — hematosis
Secondary Malignancy - possibly related to cancer treatment (Specify, __) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — skin lesion
Seizure (Nervous system disorders) | 0 | 2 | 0
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 0 | 2
Supraventricular and nodal arrhythmia - Atrial tachycardia/Paroxysmal Atrial Tachycardia (Cardiac disorders) | 0 | 0 | 1
Supraventricular and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 1 | 4
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab (N=31) | Cetuximab and Carboplatin After Cetuximab Alone (N=25) | Cetuximab and Carboplatin (N=71)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 1 | 3
Alkaline phosphatase (Investigations) | 6 | 6 | 9
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 | 0 | 5
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 1 | 1 | 5
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 | 2 | 5
Anorexia (Metabolism and nutrition disorders) | 6 | 2 | 17
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 2 | 4 | 6
Breast function/lactation (Reproductive system and breast disorders) | 0 | 0 | 2
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Injury, poisoning and procedural complications) | 1 | 0 | 1
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 0 | 4
Cardiac General - Other (Specify, __) (Cardiac disorders) | 1 | 0 | 1 — Verbatim: Edema; low blood pressure
Constipation (Gastrointestinal disorders) | 3 | 4 | 28
Constitutional Symptoms - Other (Specify, __) (General disorders) | 0 | 0 | 6 — Verbatim: performance status decrease; sinus congestion (2); heat/cold intolerance; dsyphasia; indigestion
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 21
Creatinine (Metabolism and nutrition disorders) | 0 | 0 | 2
Cystitis (Renal and urinary disorders) | 0 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 4 | 2 | 16 — Verbatim: Acne; intranasal irritation; xerosis; chelitis; hirsutism; erythema; pimple; pustules/fissures; cracked tooth; peeling cuticles; ecchymosis; ingrown toenails; skin cuts; skin sensitivity; sore thumbs; skin changes; skin cracks; dermatitis
Diarrhea (Gastrointestinal disorders) | 6 | 1 | 18
Dizziness (Nervous system disorders) | 4 | 2 | 9
Dry eye syndrome (Eye disorders) | 1 | 0 | 2
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 4 | 18
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 | 1 | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 23
Edema: limb (Blood and lymphatic system disorders) | 5 | 1 | 9
Extremity-lower (gait/walking) (General disorders) | 2 | 0 | 0
Fatigue (asthenia, lethargy, malaise) (General disorders) | 14 | 14 | 45
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3 | 2 | 3
Flushing (Vascular disorders) | 0 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 3 | 1 | 3 — Verbatim: Sore tongue; abdominal distention; indigestion; intestinal gas; heart burn; white coating in mouth
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 | 1 | 5
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 2 | 0 | 7
Heartburn/dyspepsia (Gastrointestinal disorders) | 3 | 1 | 8
Hemoglobin (Blood and lymphatic system disorders) | 2 | 2 | 13
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Hot flashes/flushes (Vascular disorders) | 6 | 1 | 12
Hypertension (Cardiac disorders) | 1 | 0 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Eye NOS (Infections and infestations) | 0 | 1 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Joint (Infections and infestations) | 1 | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 1 | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 0 | 2 | 4
Infection with normal ANC or Grade 1 or 2 neutrophils - Ungual (nails) (Infections and infestations) | 1 | 1 | 2
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 0 | 1 | 3
Infection with normal ANC or Grade 1 or 2 neutrophils - Vagina (Infections and infestations) | 1 | 0 | 1
Infection with unknown ANC - Sinus (Infections and infestations) | 0 | 1 | 1
Infection with unknown ANC - Skin (cellulitis) (Infections and infestations) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 6 | 2 | 15
Joint-function (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 0 | 1 | 9
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 5
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 | 6 | 10
Memory impairment (Nervous system disorders) | 2 | 0 | 3
Metabolic/Laboratory - Other (Specify, __) (Metabolism and nutrition disorders) | 1 | 1 | 1 — Verbatim: Increased Alkaline Phosphatase; Elevated PTT; Hematuria
Mood alteration - Anxiety (Psychiatric disorders) | 5 | 2 | 15
Mood alteration - Depression (Psychiatric disorders) | 0 | 2 | 12
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2 | 2 | 14
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 5 | 1 | 5
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 — Verbatim: Leg cramps; hand weakness; focal tenderness over the sternum; neck stiffness; sprained left ankle; stiffness
Nail changes (Skin and subcutaneous tissue disorders) | 3 | 3 | 7
Nausea (Gastrointestinal disorders) | 7 | 10 | 35
Neurology - Other (Specify, __) (Nervous system disorders) | 0 | 1 | 3 — Verbatim: gait imbalance; drooling; nightmares; tingling in legs and arms
Neuropathy: motor (Nervous system disorders) | 0 | 0 | 2
Neuropathy: sensory (Nervous system disorders) | 7 | 3 | 20
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 | 5 | 16
Ocular/Visual - Other (Specify, __) (Eye disorders) | 0 | 0 | 4 — Verbatim: Eye irritation; Left eye dropping; Bilateral Lower Eyelid Irritation; puffy right eye
Pain - Abdomen NOS (Gastrointestinal disorders) | 3 | 3 | 4
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 1 | 13
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
Pain - Breast (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Pain - Buttock (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain - Cardiac/heart (Cardiac disorders) | 0 | 1 | 2
Pain - Chest wall (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 4
Pain - Chest/thorax NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 | 4 | 4
Pain - Head/headache (Nervous system disorders) | 10 | 5 | 7
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4 | 2 | 10
Pain - Liver (Hepatobiliary disorders) | 0 | 1 | 1
Pain - Lymph node (Blood and lymphatic system disorders) | 0 | 0 | 3
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Pain - Neck (Musculoskeletal and connective tissue disorders) | 1 | 0 | 4
Pain - Other (Specify, __) (General disorders) | 8 | 4 | 10 — Verbatim: chest wall; L neck/shoulder; back; Chest pain R side w/ pleuritic component; plantar surface L foot; rib cage; R flank; pain due to acneiform rash; arm; pelvis, RUQ, L axilla; R shoulder; Right upper quadrant pain; Pain d/t Pleurex catheter
Pain - Pain NOS (General disorders) | 1 | 0 | 3
Pain - Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Platelets (Blood and lymphatic system disorders) | 0 | 2 | 14
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 | 1 | 10
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 | 2 | 7
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 — Verbatim: Wheezing; chest congestion; Upper Respiratory Infection; post nasal drip - mornings; sore throat
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 | 4 | 15
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 11 | 10 | 42
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 2 | 1 | 6
Rigors/chills (General disorders) | 1 | 0 | 1
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 1 | 1
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Taste alteration (dysgeusia) (Nervous system disorders) | 1 | 1 | 4
Tremor (Nervous system disorders) | 0 | 0 | 2
Vaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 4
Vision-blurred vision (Eye disorders) | 1 | 1 | 0
Vision-flashing lights/floaters (Eye disorders) | 1 | 0 | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5
Vomiting (Gastrointestinal disorders) | 4 | 4 | 21
Watery eye (epiphora, tearing) (Eye disorders) | 2 | 0 | 1
Weight gain (Metabolism and nutrition disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes